CLINICAL TRIAL: NCT07139392
Title: A Clinical Comparison of Connective Tissue Graft and Alb-PRF for Rebuilding Interdental Papilla
Acronym: ALB-PRF & CTG
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: shaimaa hamdy (Other)
Responsible Party: Sponsor-Investigator, shaimaa hamdy, lecturer of oral medicine, oral diagnosis and periodontology, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALB -PRF in papilla; committee 1165 (Other: ethical committee faculty of dentistry minia university)
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Papilla Reconstruction
Keywords: ALB-PRF; papilla; connective tissue; reconstruction; MINST
MeSH Terms: interventions — Albumins

STUDY DESIGN:
Intervention Model Description: Sample Selection:
  * Inclusion Criteria:
    * Age 20-55 years
    * Nordland and Tarnow Class I/II papillary loss
    * Good oral hygiene (FMPS & FMBS <20%)
    * Systemically healthy
  * Exclusion Criteria:
    * Smoking
    * Periodontal pockets >4 mm in target site
    * History of systemic diseases or medications affecting healing
    * Pregnant or lactating women
  * Preoperative Phase:
    * Oral hygiene instruction
    * Phase I periodontal therapy
    * Initial photography and papillary height measurements using digital calipers or customized stents
  * Surgical Technique:
    * Local anesthesia
    * Intrasulcular incision around target teeth
    * Papilla preservation flap
    * Harvesting CTG from the palate
    * Injection of liquid Bio-PRF at the papillary base (test group)
    * CTG positioned in the papilla region
    * Suturing with microsurgical technique
  * Postoperative Protocol:
    * Analgesics (e.g., ibuprofen 400 mg)
    * Chlorhexidine 0.12% mouth rinse for 2 weeks
    * Suture removal at 10-14 days
    * Follow-up
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- connective tissue graft (Placebo Comparator): Semi-lunar flap elevation, then connective tissue graft sutured under the flap for papilla reconstruction
  Interventions: Biological: connective tissue graft
- albumin-PRF (Active Comparator): Albumin- PRF for papilla reconstruction
  Interventions: Biological: Albumin (5% serum-protein solution containing immunoglobulins)

INTERVENTIONS:
Biological: Albumin (5% serum-protein solution containing immunoglobulins) — * Preoperative Phase:
    * Oral hygiene instruction
    * Phase I periodontal therapy
    * Initial photography and papillary height measurements using digital calipers or customized stents
  * Surgical Technique:
    * Local anesthesia
    * Intrasulcular incision around target teeth
    * Papilla preservation flap
    * Harvesting CTG from the palate
    * Injection of liquid Bio-PRF at the papillary base (test group)
    * CTG positioned in the papilla region
    * Suturing with microsurgical technique
  * Postoperative Protocol:
    * Analgesics (e.g., ibuprofen 400 mg)
    * Chlorhexidine 0.12% mouth rinse for 2 weeks
    * Suture removal at 10-14 days
    * Follow-up at 1 month, 3 months, and 6 months
  Other Names: alb-prf
  Arms: albumin-PRF
Biological: connective tissue graft — Local anesthesia. Intrasulcular incision around target teeth. Papilla preservation flap. Harvesting CTG from the palate
  Arms: connective tissue graft

SUMMARY:
The interdental papilla, a small wedge of gingival tissue positioned between adjacent teeth, plays a crucial role in both dental esthetics and oral function. Loss or deficiency of the papilla results in the formation of "black triangles," which not only compromise a patient's smile but also lead to challenges such as food impaction, phonetic difficulties, and increased risk of periodontal disease. The reconstruction of the interdental papilla is recognized as one of the most challenging procedures in periodontal therapy, particularly when aiming for enhanced esthetic outcomes and patient satisfaction

DETAILED DESCRIPTION:
Connective tissue grafts (CTG) have traditionally been regarded as the gold standard for papilla reconstruction due to their predictable augmentation of soft tissues and stable long-term results. However, CTG procedures are invasive, requiring tissue harvesting from a donor site (often the palate), and are associated with increased surgical morbidity and discomfort for patients.

Advances in regenerative medicine have introduced minimally invasive alternatives, such as injectable biologically active platelet-rich fibrin (Bio-PRF). Bio-PRF is an autologous platelet concentrate containing a high concentration of growth factors, fibrin matrix, and immunomodulatory cells. The injectable form is designed to be applied directly into tissue-deficient papillary sites, promoting enhanced angiogenesis, cell proliferation, and tissue regeneration with minimal trauma and improved patient comfort.

Recent clinical interest has focused on comparing these two approaches, CTG and injectable Bio-PRF, in their efficacy for papilla regeneration. While both techniques have demonstrated potential benefits, direct comparative studies are limited. Understanding the relative effectiveness, esthetic outcomes, surgical morbidity, and patient-centered results of these interventions is essential for evidence-based clinical decision making.

This clinical comparison seeks to evaluate and contrast the outcomes of connective tissue grafting and injectable Bio-PRF in the reconstruction of lost or compromised interdental papillae. The study aims to provide valuable insights into the optimal management of papillary defects, guiding periodontal practitioners toward treatments that maximize esthetic and functional results while minimizing patient morbidity.

We hypothesized that no significant difference between the treatment of interdental papilla with connective tissue graft or Bio-PRF.

Aim of the study

Primary Objective:

To assess the effectiveness of CTG combined with Bio-PRF in increasing papillary height in patients with papillary loss (Nordland and Tarnow Class I or II).

Secondary Objectives:

* To evaluate changes in patient satisfaction and aesthetic outcomes.
* To assess soft tissue healing and clinical attachment gain.

Materials and methods:

Study Design:

* Type: Randomized Controlled Clinical Trial
* Duration: 6 months follow-up
* Groups:

  * Group A (control): CTG alone
  * Group B (study): injectable Bio-PRF

Sample Selection:

* Inclusion Criteria:

  * Age 20-55 years
  * Nordland and Tarnow Class I/II papillary loss
  * Good oral hygiene (FMPS & FMBS <20%)
  * Systemically healthy
* Exclusion Criteria:

  * Smoking
  * Periodontal pockets >4 mm in target site
  * History of systemic diseases or medications affecting healing
  * Pregnant or lactating women
* Preoperative Phase:

  * Oral hygiene instruction
  * Phase I periodontal therapy
  * Initial photography and papillary height measurements using digital calipers or customized stents
* Surgical Technique:

  * Local anesthesia
  * Intrasulcular incision around target teeth
  * Papilla preservation flap
  * Harvesting CTG from the palate
  * Injection of liquid Bio-PRF at the papillary base (test group)
  * CTG positioned in the papilla region
  * Suturing with microsurgical technique
* Postoperative Protocol:

  * Analgesics (e.g., ibuprofen 400 mg)
  * Chlorhexidine 0.12% mouth rinse for 2 weeks
  * Suture removal at 10-14 days
  * Follow-up at 1 month, 3 months, and 6 months

Outcome Measures:

* Primary Outcome:

  o Papilla Height Gain (measured from contact point to papilla tip)
* Secondary Outcomes:

  * Visual Analog Scale (VAS) for aesthetic satisfaction
  * Healing Index
  * Black triangle area (measured via intraoral photographs or digital scanning)

Statistical Analysis:

* Descriptive statistics for baseline data
* Paired t-test or Wilcoxon signed-rank test (intragroup comparison)
* Independent t-test or Mann-Whitney U test (intergroup comparison)
* p-value < 0.05 considered statistically significant

ELIGIBILITY:
Inclusion Criteria:

* Age 20-55 years
* Nordland and Tarnow Class I/II papillary loss
* Good oral hygiene (FMPS & FMBS <20%)
* Systemically healthy

Exclusion Criteria:

* Smoking
* Periodontal pockets >4 mm in the target site
* History of systemic diseases or medications affecting healing
* Pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-09-23 (Estimated)

PRIMARY OUTCOMES:
Papilla Height Gain | 6 months follow up
  Papilla Height Gain (measured from contact point to papilla tip)

CONTACTS AND LOCATIONS:
Overall Officials: shaimaa Hamdy, lecturer, Principal Investigator — lecturer of periodontology Nahda University

IPD SHARING:
Plan to Share IPD: No
After completing the study, I will share all the data of the study

REFERENCES:
- See also: Modified interproximal tunneling technique with customized sub-epithelial connective tissue graft for gingival papilla reconstruction: report of three cases with a cutback incision on the palatal side — https://bmcoralhealth.biomedcentral.com/articles/10.1186/s12903-023-03525-7